CLINICAL TRIAL: NCT02575781
Title: A First-in-human Phase 1 Dose Escalation Study of SAR428926 in Patients With Advanced Solid Tumors
Brief Title: A Study of SAR428926 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TED14147; 2015-001441-92 (EudraCT Number); U1111-1168-4706 (Other: UTN)
Record Dates: First submitted 2015-10-08; First posted 2015-10-15 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Neoplasm Malignant
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- SAR428926-Escalating cohort (Experimental): SAR428926 will be administered intravenously up to disease progression or dose limiting toxicities
  Interventions: Drug: SAR428926
- SAR428926 in triple negative breast cancer-Expansion Cohort 1 (Experimental): SAR428926 will be administered intravenously at maximum tolerated dose (MTD) up to disease progression or unacceptable toxicity
  Interventions: Drug: SAR428926
- SAR428926 in solid tumors-Expansion Cohort 2 (Experimental): SAR428926 will be administered intravenously at the MTD up to disease progression or unacceptable toxicity
  Interventions: Drug: SAR428926

INTERVENTIONS:
Drug: SAR428926 — Pharmaceutical form:concentrate for solution for infusion Route of administration: intravenous

SUMMARY:
Primary Objectives:

To determine the maximum tolerated dose (MTD) of SAR428926 when administered as a single agent in patients with advanced solid tumors.

To evaluate the anti-tumor response of SAR428926 when administered as a single agent in patients with advanced triple negative breast cancer (TNBC) positive for the protein targeted by SAR428926 To assess the preliminary anti-tumor response of SAR428926 when administered as a single agent in patients with advanced solid tumors positive for the protein targeted by SAR428926

Secondary Objectives:

To determine the overall safety profile of SAR428926 as a single agent. To characterize the pharmacokinetics (PK) profile of SAR428926 and its metabolites.

To identify the recommended Phase 2 dose (RP2D) of SAR428926 as a single agent. To evaluate the immunogenicity of SAR428926. To assess the tumor response and duration of tumor response in all treated patients.

To evaluate the benefit of primary prophylaxis on the occurrence of corneal (keratopathy/keratitis) toxicity (Expansion cohorts).

DETAILED DESCRIPTION:
The study duration for an individual patient will include a screening period for inclusion of up to 28 days, a treatment period, an end-of-treatment (EOT) visit around 30 days following the last administration of SAR428926, and at least one follow-up visit around 30 days after the EOT visit. The treatment period may continue until disease progression, intolerable toxicity, or investigator, Sponsor, or patient decision to discontinue therapy. Patients who discontinue treatment for reasons other than progression of disease will be followed every 3 months until progression, initiation of subsequent therapy, or until the primary analysis cutoff date, whichever comes first.

ELIGIBILITY:
Inclusion criteria :

* Patients with advanced solid tumor with no standard alternative treatment.
* Availability of archived tumor tissue for SAR428926 targeted antigen testing.
* For participants in the Escalation Phase: human epidermal growth factor receptor 2 (HER2) negative breast cancer (BC), gastric cancer, colorectal cancer (CRC), ovarian cancer, prostate cancer and non small-cell lung cancer (NSCLC).
* For participants in the Expansion Phase: patients with TNBC, prostate cancer, CRC, ovarian cancer or NSCLC and positive SAR428926 targeted antigen.
* At least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and one lesion amenable to biopsy in expansion cohort only (except for NSCLC patients).

Exclusion criteria:

* Age less than 18 years old.
* Eastern Cooperative Oncology Group (ECOG) performance status more than 1.
* New or progressing brain metastases.
* Concurrent treatment with any other anticancer therapy or inadequate wash-out period for prior anticancer therapies, including other experimental anticancer treatment, before first administration of SAR428926, or non resolution of toxicities induced by these anticancer therapies.
* Women of reproductive potential and male subjects with female partners of childbearing potential who are not willing to avoid pregnancy.
* Pregnancy or breast feeding.
* Prior maytansinoid treatments (DM1 or DM4 antibody drug conjugates [ADCs]).
* Unwillingness and inability to comply with scheduled visits, drug administration plan, laboratory tests, other study procedures, and study restrictions.
* Significant concomitant illness, including psychiatric condition that, in the opinion of the Investigator or Sponsor, would adversely affect the patient's participation in the study.
* Any surgery within the preceding 3 weeks.
* Known human immunodeficiency virus (HIV) infection or active hepatitis B or C viral infection.
* Poor bone marrow reserve.
* Poor kidney and liver function.
* Previous history of chronic corneal diseases (even if asymptomatic) or unresolved acute non-recurrent corneal conditions. Patients wearing contact lenses who are not willing to stop wearing them for the duration of the study.
* Unresolved signs and symptoms of peripheral neuropathy; Grade 1 is acceptable.
* Abnormal cardiac function defined by a left ventricular ejection fraction (LVEF) <50%.
* Known intolerance to infused protein products including other monoclonal antibodies and ADCs.
* Medical conditions requiring concomitant administration of medications with narrow therapeutic window, metabolized by CYPs and which a dose reduction cannot be considered.
* Medical conditions requiring concomitant administration of strong CYP3A inhibitors, unless it can be discontinued at least two weeks before first administration of SAR428926.
* Other prior neoplasm.
* Contraindications to the use of ophthalmic vasoconstrictor and/or corticosteroid as per package insert of each drug, including the following: increase intraocular pressure, prior or current glaucoma, narrow-angle glaucoma, ongoing eye infection, uncontrolled hypertension, known/suspected allergy to constituents of the preparation (such as sodium bisulfite).

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-10-05 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Number of patients with dose limiting adverse events (Escalation cohort) | 4 weeks
Number of patients with corneal adverse events impacting study treatment (Escalation cohort) | 8 weeks
Assessment of overall response rate using standard imaging and RECIST v1.1 criteria (Expansion cohort) | Tumor assessment every 2 months until disease progression or up to 36 months, whichever came first

SECONDARY OUTCOMES:
Number of treatment emergent adverse events | Up to 3 years
Assessment of PK parameter: maximum concentration (Cmax) | 2 months
Assessment of PK parameter: time to reach maximum concentration (tmax) | 2 months
Assessment of PK parameter: trough plasma concentration (Ctrough) | Every 2 weeks until approximately 14 weeks
Assessment of PK parameter: area under the plasma concentration curve versus time curve between 1 and 14 days (AUC0-14 day) | 2 months
Assessment of PK parameter: mean systemic clearance (CL) | 2 months
Assessment of PK parameter: clearance at steady state (CLss) | 2 months
Assessment of PK parameter: accumulation ratio on AUC0-14 | 2 months
Assessment of PK parameter: accumulation ratio on Cmax | 2 months
Preliminary tumor response by RECIST v1.1 (Escalation) | 2 months
Number of corneal events according to the presence or not of preventive measures | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (3):
- Investigational Site Number 2080001, København Ø, Denmark
- Investigational Site Number 2500001, Villejuif, France
- Investigational Site Number 7240001, Barcelona, Spain